CLINICAL TRIAL: NCT05630339
Title: Efficacy and Security of the Magnesium and Vitamin D Combination as Adjuvant Treatment of Post-COVID Syndrome. A Randomised Double-blind Clinical Trial
Brief Title: Magnesium and Vitamin D Combination for Post-COVID Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Consejo de Ciencia y Tecnología del Estado de Durango (Unknown)
Responsible Party: Principal Investigator, Fernando Guerrero Romero MD, Director of the research unit, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R-2021-785-076
Record Dates: First submitted 2022-11-08; First posted 2022-11-29 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Post-COVID-19 Syndrome; Long COVID; Vitamin D Deficiency; Magnesium Deficiency
Keywords: Post-COVID syndrome; Long COVID; Vitamin D; Magnesium
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Vitamin D Deficiency; Magnesium Deficiency | interventions — Magnesium Chloride; Magnesium; Vitamin D; Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Study groups:
  1. Intervention group that will receive 1.2 g of magnesium chloride (equivalent to 360 mg of magnesium elemental) + 4000 IU of vitamin D once a day, for four months.
  2. Control group that will receive inert placebo for four months.
Who Masked: Participant, Care Provider
Masking Description: Neither the patient nor the treating doctor will know the study group the participant was randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Will receive 1.2 g of magnesium chloride (equivalent to 360 mg of magnesium elemental) + 4000 IU of vitamin D once a day, for four months.
  Interventions: Dietary Supplement: Magnesium chloride; Dietary Supplement: Vitamin D
- Control group. (Placebo Comparator): Will receive inert placebo for four months.
  Interventions: Dietary Supplement: Inert placebo

INTERVENTIONS:
Dietary Supplement: Magnesium chloride — Each 650 mg capsule contains 340 mg of magnesium chloride, which must be ingested twice a day with aliments.
  Other Names: Magnesium
  Arms: Intervention group
Dietary Supplement: Vitamin D — Each tablet contains 4000 IU of vitamin D, and must be ingested a pill per night.
  Other Names: Cholecalciferol
  Arms: Intervention group
Dietary Supplement: Inert placebo — Instead of dietary supplements, sodium bicarbonate as inert placebo will be administered twice a day in 650 mg capsules.
  Arms: Control group.

SUMMARY:
The goal of this double-blind randomized controlled clinical trial is to determine the efficacy of the administration of magnesium chloride + vitamin D as an adjuvant in the treatment of post-Coronavirus Disease (COVID) syndrome.

The participants will be integrated: a) Intervention group that will receive 1 g of magnesium chloride (equivalent to 300 mg of elemental magnesium) + 4000 IU of vitamin D once a day, for four months. b) Control group that will receive inert placebo for four months.

The outcome variable will be the improvement of the post-COVID syndrome. At the beginning and end of the study, blood samples will be taken to determine serum levels of vitamin D, total magnesium, ionic magnesium, calcium, fasting glucose and lipid profile.

The evaluation of the efficacy and safety of the proposed intervention will be carried out by establishing the differences between the intervention and control groups.

DETAILED DESCRIPTION:
More than 50 signs and symptoms have been described that characterize the post-COVID syndrome, among them the early presence of fatigue, shortness of breath, cough, joint and chest pain. Later, the signs and symptoms that may occur are muscle pain, headache, tachycardia, loss of smell or taste, memory and concentration problems, difficulty falling asleep, skin rashes and hair loss.

Vitamin D is a fat-soluble vitamin whose best-known function is calcium and phosphate homeostasis, but it is also involved in multiple processes, including the regulation of the immune response. In vitro, vitamin D decreases viral replication, which is linked to its ability to stimulate innate immunity, increases the synthesis of cathelicidin and defensins, peptides that favor the preservation of the mucosa and enhance its protective effect against infection. In vivo, vitamin D decreases the expression of the cellular co-receptor dipeptidyl peptidase (DPP)-4/cluster of differentiation antigen 26 (CD26), which interacts with protein S, which decreases the penetration of the virus into the cell, contributes to the regulation of immunity, regulating excessive immune response, which is associated with an adverse prognosis, and interacts with the nuclear factor-kappa B (NF-kB) pathway, decreases the intensity of the Th1 response and the synthesis of proinflammatory cytokines, and increases the synthesis of anti-inflammatory cytokines.

Magnesium, through its calcium channel blocking effect, decreases the inflammatory response produced by the NF-kB cascade, reduces the production of tumor necrosis factor alpha (TNF-α) and interleukin 6 (IL-6) by monocytes and the expression of cytokines and inflammatory proteins. It influences both cell-mediated and humoral adaptive immunity, since it participates in the activation of leukocytes, the binding of antigens to macrophages, apoptotic regulation, and it reduces the production of superoxide anions.

The pathophysiology of the post-COVID syndrome is not precisely known, although it has been established that it is a disorder with inflammatory components, endothelial damage, and thromboembolism.

In this context, magnesium deficiency is associated with the development of the pro-inflammatory and pro-thrombotic response that generates a favorable microenvironment for the development of inflammation, endothelial damage and thromboembolism, components linked to the post-COVID syndrome. On the other hand, it has been described that patients with post-COVID present with vitamin D deficiency, a deficiency that contributes to the development of fatigue, anemia and chronic inflammation. In addition, there is interaction between magnesium and vitamin D, in such a way that the deficiency of the first contributes to the decrease in the synthesis of 25-hydroxy vitamin D and 1,25-hydroxy vitamin D and the number and activity of vitamin D receptors.

Therefore, it is plausible to assume that both magnesium and vitamin D play an important role in the development of post-COVID syndrome.

Goal. To determine the efficacy of the administration of magnesium chloride + vitamin D as an adjuvant in the treatment of post-COVID syndrome.

Methods. Double-blind randomized controlled clinical trial to which subjects diagnosed with post-COVID syndrome will be integrated. The participants will be integrated: a) Intervention group that will receive 1 g of magnesium chloride (equivalent to 300 mg of elemental magnesium) + 4000 IU of vitamin D once a day, for four months. b) Control group that will receive inert placebo for four months.

Men and women, aged 18 years or older, with a diagnosis of post-COVID syndrome, hypomagnesaemia and vitamin D insufficiency will be included. Having received magnesium or vitamin D supplements in the last 30 days, as well as treatment based on of steroids, will be exclusion criteria. The withdrawal of informed consent and adherence to the intervention less than 80% will be criteria for elimination.

The outcome variable will be the improvement of the post-COVID syndrome. At the beginning and end of the study, blood samples will be taken to determine serum levels of vitamin D, total magnesium, ionic magnesium, calcium, fasting glucose and lipid profile.

Statistic analysis. The evaluation of the efficacy and safety of the proposed intervention will be carried out by establishing the differences between the intervention and control groups, which will be estimated using the unpaired Student's t-test for analysis of the parametric variables (Mann-Whitney U for non-parametric variables) and Chi-Square (Fisher's exact test) for the analysis of categorical variables.

Intragroup differences will be estimated using the paired Student's t-test. Even when it is assumed that the confounding variables will be controlled by the randomization process; Additionally, a stratified analysis will be carried out by those confounding variables that in the bivariate analysis show significant differences.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 or older.
* Previous diagnosis of COVID-19, confirmed by Real Time Polymerase Chain Reaction (RT-PCR) for Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2)
* Diagnosis of post-COVID syndrome
* Hypomagnesemia
* Vitamin D deficiency

Exclusion Criteria:

* Subjects who have received magnesium and/or vitamin D supplements in the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Post-COVID syndrome symptoms at 4 months | First control date, and four months after treatment initiation.
  The presence of two or more of the following signs and/or symptoms will be considered a suspicion of post-COVID syndrome: Fatigue, shortness of breath, cough, joint pain, chest pain, muscle pain, headache, tachycardia, arrhythmias, loss of smell, loss of taste, memory problems, concentration problems, depression, anxiety, insomnia, skin rashes, hair loss.
Change from Baseline Post-COVID Functional Status at 4 months | First control date, and four months after treatment initiation.
  Post-COVID Functional Status Scale
Change from Baseline Serum vitamin D levels at 4 months | First control assessment, and four months after treatment initiation.
  Recovery of serum vitamin D levels from deficiency (< 30 ng/mL) to normally (30 - 100 ng/mL).
  The serum concentration of the 25 OH vitamin D fraction will be determined by the enzyme-linked immunosorbent assay (ELISA) method, the serum levels of magnesium and calcium by colorimetric techniques (A15 Clinical Analyzer, Biosystems, USA).
Change from Baseline Serum Magnesium levels at 4 months | First control assessment, and four months after treatment initiation.
  Recovery of serum magnesium levels from deficiency (< 2.0 mg/dL) to normally (2.0 - 2.5 mg/dL).
Change from Baseline Mental State levels at 4 months | First control date, and four months after treatment initiation.
  Mini Mental State Examination
Change from Baseline Anxiety Symptoms at 4 months | First control date, and four months after treatment initiation.
  Beck Anxiety Inventory
Change from Baseline Depression Symptoms at 4 months | First control date, and four months after treatment initiation.
  Beck Depression Inventory
Change from Baseline Post-traumatic Stress Symptoms at 4 months | First control date, and four months after treatment initiation.
  Severity of Post-traumatic Stress Symptoms
Change from Baseline Dyspnea Symptoms at 4 months | First control date, and four months after treatment initiation.
  modified Medical Research Council (mMRC) dyspnea scale

SECONDARY OUTCOMES:
Change from Baseline Fasting Blood Glucose levels at 4 months | First control assessment, and four months after treatment initiation.
  Normal values: 70 - 100 mg/dL
Change from Baseline Serum Lipid Profile at 4 months | First control assessment, and four months after treatment initiation.
  Normal values: total cholesterol 100 - 200 mg/dL; HDL-cholesterol 40 - 60 mg/dL; triglycerides 50 - 150 mg/dL.
Change from Baseline Serum Calcium levels at 4 months | First control assessment, and four months after treatment initiation.
  Normal values: 8.4 - 10.2 mg/dL
Change from Baseline Serum Creatinine levels at 4 months | First control assessment, and four months after treatment initiation.
  Normal values: 0.5 - 1.2 mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Guerrero, PhD, Principal Investigator — Instituto Mexicano del Seguro Social; Gerardo Martínez, PhD, Study Chair — Instituto Mexicano del Seguro Social; Luis Simental, PhD, Study Chair — Instituto Mexicano del Seguro Social
Locations (1):
- Biomedical Research Unit. IMSS. Durango, Durango, Durango, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ackermann M, Verleden SE, Kuehnel M, Haverich A, Welte T, Laenger F, Vanstapel A, Werlein C, Stark H, Tzankov A, Li WW, Li VW, Mentzer SJ, Jonigk D. Pulmonary Vascular Endothelialitis, Thrombosis, and Angiogenesis in Covid-19. N Engl J Med. 2020 Jul 9;383(2):120-128. doi: 10.1056/NEJMoa2015432. Epub 2020 May 21. PMID 32437596
- [Background] Addison AB, Wong B, Ahmed T, Macchi A, Konstantinidis I, Huart C, Frasnelli J, Fjaeldstad AW, Ramakrishnan VR, Rombaux P, Whitcroft KL, Holbrook EH, Poletti SC, Hsieh JW, Landis BN, Boardman J, Welge-Lussen A, Maru D, Hummel T, Philpott CM. Clinical Olfactory Working Group consensus statement on the treatment of postinfectious olfactory dysfunction. J Allergy Clin Immunol. 2021 May;147(5):1704-1719. doi: 10.1016/j.jaci.2020.12.641. Epub 2021 Jan 13. PMID 33453291
- [Background] Ali N. Role of vitamin D in preventing of COVID-19 infection, progression and severity. J Infect Public Health. 2020 Oct;13(10):1373-1380. doi: 10.1016/j.jiph.2020.06.021. Epub 2020 Jun 20. PMID 32605780
- [Background] Amenta EM, Spallone A, Rodriguez-Barradas MC, El Sahly HM, Atmar RL, Kulkarni PA. Postacute COVID-19: An Overview and Approach to Classification. Open Forum Infect Dis. 2020 Oct 21;7(12):ofaa509. doi: 10.1093/ofid/ofaa509. eCollection 2020 Dec. PMID 33403218
- [Background] Aranow C. Vitamin D and the immune system. J Investig Med. 2011 Aug;59(6):881-6. doi: 10.2310/JIM.0b013e31821b8755. PMID 21527855
- [Background] Becker RC. COVID-19 and its sequelae: a platform for optimal patient care, discovery and training. J Thromb Thrombolysis. 2021 Apr;51(3):587-594. doi: 10.1007/s11239-021-02375-w. Epub 2021 Jan 27. PMID 33501596
- [Background] Behl T, Kaur I, Bungau S, Kumar A, Uddin MS, Kumar C, Pal G, Sahil, Shrivastava K, Zengin G, Arora S. The dual impact of ACE2 in COVID-19 and ironical actions in geriatrics and pediatrics with possible therapeutic solutions. Life Sci. 2020 Sep 15;257:118075. doi: 10.1016/j.lfs.2020.118075. Epub 2020 Jul 10. PMID 32653522
- [Background] Bellan M, Soddu D, Balbo PE, Baricich A, Zeppegno P, Avanzi GC, Baldon G, Bartolomei G, Battaglia M, Battistini S, Binda V, Borg M, Cantaluppi V, Castello LM, Clivati E, Cisari C, Costanzo M, Croce A, Cuneo D, De Benedittis C, De Vecchi S, Feggi A, Gai M, Gambaro E, Gattoni E, Gramaglia C, Grisafi L, Guerriero C, Hayden E, Jona A, Invernizzi M, Lorenzini L, Loreti L, Martelli M, Marzullo P, Matino E, Panero A, Parachini E, Patrucco F, Patti G, Pirovano A, Prosperini P, Quaglino R, Rigamonti C, Sainaghi PP, Vecchi C, Zecca E, Pirisi M. Respiratory and Psychophysical Sequelae Among Patients With COVID-19 Four Months After Hospital Discharge. JAMA Netw Open. 2021 Jan 4;4(1):e2036142. doi: 10.1001/jamanetworkopen.2020.36142. PMID 33502487
- [Background] Britton J, Pavord I, Richards K, Wisniewski A, Knox A, Lewis S, Tattersfield A, Weiss S. Dietary magnesium, lung function, wheezing, and airway hyperreactivity in a random adult population sample. Lancet. 1994 Aug 6;344(8919):357-62. doi: 10.1016/s0140-6736(94)91399-4. PMID 7914305
- [Background] Carvalho-Schneider C, Laurent E, Lemaignen A, Beaufils E, Bourbao-Tournois C, Laribi S, Flament T, Ferreira-Maldent N, Bruyere F, Stefic K, Gaudy-Graffin C, Grammatico-Guillon L, Bernard L. Follow-up of adults with noncritical COVID-19 two months after symptom onset. Clin Microbiol Infect. 2021 Feb;27(2):258-263. doi: 10.1016/j.cmi.2020.09.052. Epub 2020 Oct 5. PMID 33031948
- [Background] Dennis A, Wamil M, Alberts J, Oben J, Cuthbertson DJ, Wootton D, Crooks M, Gabbay M, Brady M, Hishmeh L, Attree E, Heightman M, Banerjee R, Banerjee A; COVERSCAN study investigators. Multiorgan impairment in low-risk individuals with post-COVID-19 syndrome: a prospective, community-based study. BMJ Open. 2021 Mar 30;11(3):e048391. doi: 10.1136/bmjopen-2020-048391. PMID 33785495
- [Background] Garg P, Arora U, Kumar A, Malhotra A, Kumar S, Garg S, Arora M, Sarda R, Wig N. Risk factors for prolonged fatigue after recovery from COVID-19. J Med Virol. 2021 Apr;93(4):1926-1928. doi: 10.1002/jmv.26774. Epub 2021 Jan 12. No abstract available. PMID 33393696
- [Background] Gasmi A, Tippairote T, Mujawdiya PK, Peana M, Menzel A, Dadar M, Gasmi Benahmed A, Bjorklund G. Micronutrients as immunomodulatory tools for COVID-19 management. Clin Immunol. 2020 Nov;220:108545. doi: 10.1016/j.clim.2020.108545. Epub 2020 Jul 22. PMID 32710937
- [Background] Gattinoni L, Chiumello D, Caironi P, Busana M, Romitti F, Brazzi L, Camporota L. COVID-19 pneumonia: different respiratory treatments for different phenotypes? Intensive Care Med. 2020 Jun;46(6):1099-1102. doi: 10.1007/s00134-020-06033-2. Epub 2020 Apr 14. No abstract available. PMID 32291463
- [Background] Glasdam SM, Glasdam S, Peters GH. The Importance of Magnesium in the Human Body: A Systematic Literature Review. Adv Clin Chem. 2016;73:169-93. doi: 10.1016/bs.acc.2015.10.002. Epub 2016 Jan 13. PMID 26975973
- [Background] Gombart AF. The vitamin D-antimicrobial peptide pathway and its role in protection against infection. Future Microbiol. 2009 Nov;4(9):1151-65. doi: 10.2217/fmb.09.87. PMID 19895218
- [Background] Gonzalez EP, Santos F, Coto E. [Magnesium homeostasis. Etiopathogeny, clinical diagnosis and treatment of hypomagnesaemia. A case study]. Nefrologia. 2009;29(6):518-24. doi: 10.3265/Nefrologia.2009.29.6.5534.en.full. Spanish. PMID 19935995
- [Background] Grant WB, Lahore H, McDonnell SL, Baggerly CA, French CB, Aliano JL, Bhattoa HP. Evidence that Vitamin D Supplementation Could Reduce Risk of Influenza and COVID-19 Infections and Deaths. Nutrients. 2020 Apr 2;12(4):988. doi: 10.3390/nu12040988. PMID 32252338
- [Background] Greenhalgh T, Knight M, A'Court C, Buxton M, Husain L. Management of post-acute covid-19 in primary care. BMJ. 2020 Aug 11;370:m3026. doi: 10.1136/bmj.m3026. No abstract available. PMID 32784198
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Havervall S, Rosell A, Phillipson M, Mangsbo SM, Nilsson P, Hober S, Thalin C. Symptoms and Functional Impairment Assessed 8 Months After Mild COVID-19 Among Health Care Workers. JAMA. 2021 May 18;325(19):2015-2016. doi: 10.1001/jama.2021.5612. PMID 33825846
- [Background] Iotti S, Wolf F, Mazur A, Maier JA. The COVID-19 pandemic: is there a role for magnesium? Hypotheses and perspectives. Magnes Res. 2020 May 1;33(2):21-27. doi: 10.1684/mrh.2020.0465. PMID 32554340
- [Background] Jolliffe DA, Camargo CA Jr, Sluyter JD, Aglipay M, Aloia JF, Ganmaa D, Bergman P, Borzutzky A, Damsgaard CT, Dubnov-Raz G, Esposito S, Gilham C, Ginde AA, Golan-Tripto I, Goodall EC, Grant CC, Griffiths CJ, Hibbs AM, Janssens W, Khadilkar AV, Laaksi I, Lee MT, Loeb M, Maguire JL, Majak P, Mauger DT, Manaseki-Holland S, Murdoch DR, Nakashima A, Neale RE, Pham H, Rake C, Rees JR, Rosendahl J, Scragg R, Shah D, Shimizu Y, Simpson-Yap S, Kumar GT, Urashima M, Martineau AR. Vitamin D supplementation to prevent acute respiratory infections: systematic review and meta-analysis of aggregate data from randomised controlled trials. medRxiv [Preprint]. 2020 Nov 25:2020.07.14.20152728. doi: 10.1101/2020.07.14.20152728. PMID 33269357
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306
- [Background] Leta V, Rodriguez-Violante M, Abundes A, Rukavina K, Teo JT, Falup-Pecurariu C, Irincu L, Rota S, Bhidayasiri R, Storch A, Odin P, Antonini A, Ray Chaudhuri K. Parkinson's Disease and Post-COVID-19 Syndrome: The Parkinson's Long-COVID Spectrum. Mov Disord. 2021 Jun;36(6):1287-1289. doi: 10.1002/mds.28622. Epub 2021 Apr 28. No abstract available. PMID 33890344
- [Background] Liu K, Chen Y, Lin R, Han K. Clinical features of COVID-19 in elderly patients: A comparison with young and middle-aged patients. J Infect. 2020 Jun;80(6):e14-e18. doi: 10.1016/j.jinf.2020.03.005. Epub 2020 Mar 27. PMID 32171866
- [Background] Malek Mahdavi A. A brief review of interplay between vitamin D and angiotensin-converting enzyme 2: Implications for a potential treatment for COVID-19. Rev Med Virol. 2020 Sep;30(5):e2119. doi: 10.1002/rmv.2119. Epub 2020 Jun 25. PMID 32584474
- [Background] Malihi Z, Wu Z, Lawes CMM, Scragg R. Adverse events from large dose vitamin D supplementation taken for one year or longer. J Steroid Biochem Mol Biol. 2019 Apr;188:29-37. doi: 10.1016/j.jsbmb.2018.12.002. Epub 2018 Dec 6. PMID 30529281
- [Background] Maltezou HC, Pavli A, Tsakris A. Post-COVID Syndrome: An Insight on Its Pathogenesis. Vaccines (Basel). 2021 May 12;9(5):497. doi: 10.3390/vaccines9050497. PMID 34066007
- [Background] Marini JJ, Gattinoni L. Management of COVID-19 Respiratory Distress. JAMA. 2020 Jun 9;323(22):2329-2330. doi: 10.1001/jama.2020.6825. No abstract available. PMID 32329799
- [Background] Martinez-Zavala N, Lopez-Sanchez GN, Vergara-Lopez A, Chavez-Tapia NC, Uribe M, Nuno-Lambarri N. Vitamin D deficiency in Mexicans have a high prevalence: a cross-sectional analysis of the patients from the Centro Medico Nacional 20 de Noviembre. Arch Osteoporos. 2020 Jun 16;15(1):88. doi: 10.1007/s11657-020-00765-w. PMID 32542548
- [Background] Mejia-Rodriguez F, Shamah-Levy T, Villalpando S, Garcia-Guerra A, Mendez-Gomez Humaran I. Iron, zinc, copper and magnesium deficiencies in Mexican adults from the National Health and Nutrition Survey 2006. Salud Publica Mex. 2013 May-Jun;55(3):275-84. doi: 10.21149/spm.v55i3.7210. PMID 23912540
- [Background] Nielsen FH. Magnesium, inflammation, and obesity in chronic disease. Nutr Rev. 2010 Jun;68(6):333-40. doi: 10.1111/j.1753-4887.2010.00293.x. PMID 20536778
- [Background] Perez T, Burgel PR, Paillasseur JL, Caillaud D, Deslee G, Chanez P, Roche N; INITIATIVES BPCO Scientific Committee. Modified Medical Research Council scale vs Baseline Dyspnea Index to evaluate dyspnea in chronic obstructive pulmonary disease. Int J Chron Obstruct Pulmon Dis. 2015 Aug 18;10:1663-72. doi: 10.2147/COPD.S82408. eCollection 2015. PMID 26316740
- [Background] Raahimi MM, Kane A, Moore CE, Alareed AW. Late onset of Guillain-Barre syndrome following SARS-CoV-2 infection: part of 'long COVID-19 syndrome'? BMJ Case Rep. 2021 Jan 18;14(1):e240178. doi: 10.1136/bcr-2020-240178. PMID 33462068
- [Background] Rivera-Paredez B, Hidalgo-Bravo A, de la Cruz-Montoya A, Martinez-Aguilar MM, Ramirez-Salazar EG, Flores M, Quezada-Sanchez AD, Ramirez-Palacios P, Cid M, Martinez-Hernandez A, Orozco L, Denova-Gutierrez E, Salmeron J, Velazquez-Cruz R. Association between vitamin D deficiency and common variants of Vitamin D binding protein gene among Mexican Mestizo and indigenous postmenopausal women. J Endocrinol Invest. 2020 Jul;43(7):935-946. doi: 10.1007/s40618-019-01177-5. Epub 2020 Jan 6. PMID 31907821
- [Background] Rosanoff A, West C, Elin RJ, Micke O, Baniasadi S, Barbagallo M, Campbell E, Cheng FC, Costello RB, Gamboa-Gomez C, Guerrero-Romero F, Gletsu-Miller N, von Ehrlich B, Iotti S, Kahe K, Kim DJ, Kisters K, Kolisek M, Kraus A, Maier JA, Maj-Zurawska M, Merolle L, Nechifor M, Pourdowlat G, Shechter M, Song Y, Teoh YP, Touyz RM, Wallace TC, Yokota K, Wolf F; MaGNet Global Magnesium Project (MaGNet). Recommendation on an updated standardization of serum magnesium reference ranges. Eur J Nutr. 2022 Oct;61(7):3697-3706. doi: 10.1007/s00394-022-02916-w. Epub 2022 Jun 10. PMID 35689124
- [Background] Scoppettuolo P, Borrelli S, Naeije G. Neurological involvement in SARS-CoV-2 infection: A clinical systematic review. Brain Behav Immun Health. 2020 May;5:100094. doi: 10.1016/j.bbih.2020.100094. Epub 2020 Jun 6. PMID 33521692
- [Background] Shereen MA, Khan S, Kazmi A, Bashir N, Siddique R. COVID-19 infection: Origin, transmission, and characteristics of human coronaviruses. J Adv Res. 2020 Mar 16;24:91-98. doi: 10.1016/j.jare.2020.03.005. eCollection 2020 Jul. PMID 32257431
- [Background] Simani L, Ramezani M, Darazam IA, Sagharichi M, Aalipour MA, Ghorbani F, Pakdaman H. Prevalence and correlates of chronic fatigue syndrome and post-traumatic stress disorder after the outbreak of the COVID-19. J Neurovirol. 2021 Feb;27(1):154-159. doi: 10.1007/s13365-021-00949-1. Epub 2021 Feb 2. PMID 33528827
- [Background] Simental-Mendia LE, Sahebkar A, Rodriguez-Moran M, Guerrero-Romero F. A systematic review and meta-analysis of randomized controlled trials on the effects of magnesium supplementation on insulin sensitivity and glucose control. Pharmacol Res. 2016 Sep;111:272-282. doi: 10.1016/j.phrs.2016.06.019. Epub 2016 Jun 18. PMID 27329332
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Talavera JO, Rivas-Ruiz R, Bernal-Rosales LP. [Clinical research V. Sample size]. Rev Med Inst Mex Seguro Soc. 2011 Sep-Oct;49(5):517-22. Spanish. PMID 22185853
- [Background] Tan CW, Ho LP, Kalimuddin S, Cherng BPZ, Teh YE, Thien SY, Wong HM, Tern PJW, Chandran M, Chay JWM, Nagarajan C, Sultana R, Low JGH, Ng HJ. Cohort study to evaluate the effect of vitamin D, magnesium, and vitamin B12 in combination on progression to severe outcomes in older patients with coronavirus (COVID-19). Nutrition. 2020 Nov-Dec;79-80:111017. doi: 10.1016/j.nut.2020.111017. Epub 2020 Sep 8. PMID 33039952
- [Background] Uwitonze AM, Razzaque MS. Role of Magnesium in Vitamin D Activation and Function. J Am Osteopath Assoc. 2018 Mar 1;118(3):181-189. doi: 10.7556/jaoa.2018.037. PMID 29480918
- [Background] Volpe SL. Magnesium in disease prevention and overall health. Adv Nutr. 2013 May 1;4(3):378S-83S. doi: 10.3945/an.112.003483. PMID 23674807
- [Background] Weng J, Li Y, Li J, Shen L, Zhu L, Liang Y, Lin X, Jiao N, Cheng S, Huang Y, Zou Y, Yan G, Zhu R, Lan P. Gastrointestinal sequelae 90 days after discharge for COVID-19. Lancet Gastroenterol Hepatol. 2021 May;6(5):344-346. doi: 10.1016/S2468-1253(21)00076-5. Epub 2021 Mar 10. No abstract available. PMID 33711290
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] Xu J, Yang J, Chen J, Luo Q, Zhang Q, Zhang H. Vitamin D alleviates lipopolysaccharide-induced acute lung injury via regulation of the renin-angiotensin system. Mol Med Rep. 2017 Nov;16(5):7432-7438. doi: 10.3892/mmr.2017.7546. Epub 2017 Sep 20. PMID 28944831
- [Background] Xu Y, Baylink DJ, Chen CS, Reeves ME, Xiao J, Lacy C, Lau E, Cao H. The importance of vitamin d metabolism as a potential prophylactic, immunoregulatory and neuroprotective treatment for COVID-19. J Transl Med. 2020 Aug 26;18(1):322. doi: 10.1186/s12967-020-02488-5. PMID 32847594
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Result] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- See also: Patient-Led Research Collaborative. Report: What Does COVID-19 Recovery Actually Look Like? An Analysis of the Prolonged COVID-19 Symptoms Survey by Patient-Led Research Team — http://patientresearchcovid19.com/research/report-1/